CLINICAL TRIAL: NCT05230628
Title: The Effectiveness of Transcutaneous Electrical Nerve Stimulation of the Auricular Branch of the Vagus Nerve in Loss Weight and Improving the Quality of Life in Patients With Obesity
Brief Title: Auricular Vagus Stimulation in Obesity
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Medical Research Center for Therapy and Preventive Medicine (Other Government)
Collaborators: Moscow State University of Medicine and Dentistry (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 01-04/22
Record Dates: First submitted 2022-01-28; First posted 2022-02-09 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Vagus Nerve Stimulation; Obesity
Keywords: auricular stimulation; auricular vagus nerve stimulation; blinding (masking); transcutaneous vagus nerve stimulation (TENS); vagus nerve stimulation (VNS); obesity abdominal; nutrition disorders; overweight; body weight; active TENS; sham TENS; heart rate; total fat; body mass index; waist circumference; hip circumference; Heart rate variability; quality of life
MeSH Terms: conditions — Obesity; Obesity, Abdominal; Nutrition Disorders; Overweight; Body Weight

STUDY DESIGN:
Intervention Model Description: Model: 1:1 randomization of active stimulation vs. no stimulation for 6 months post randomization.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active TENS (Experimental): Active will be performed with using a TENS device with an ear clip attached to the tragus of the right ear (which is innervated by auricular branch of the vagus nerve) at 25 Hz, 200ms at a current just below discomfort threshold.
  Interventions: Device: Active TENS
- Sham TENS (Sham Comparator): Sham TENS will be performed to the ear lobe, which is devoid of vagal innervation.
  Interventions: Device: Sham TENS

INTERVENTIONS:
Device: Active TENS — Active TENS stimulation will occur daily for 10 minutes, 3-4 times a day, 30 minutes before the main meals. The duration will be 6 months for each patient.
  Arms: Active TENS
Device: Sham TENS — Sham TENS stimulation will occur daily for 10 minutes, 3-4 times a day, 30 minutes before the main meals. The duration will be 6 months for each patient.
  Arms: Sham TENS

SUMMARY:
Transcutaneous vagus nerve stimulation (TENS) involves stimulation of the left and/or right auricular branch of the vagus nerve with low-frequency electrical impulses. In recent years, the possibilities of using this technology in chronic conditions characterized by immune and metabolic dysregulation have been studied. The aim of this study is to investigate the effectiveness of TENS in reducing weight and improving quality of life in patients with various degrees of obesity.

DETAILED DESCRIPTION:
Obesity is one of the leading causes of disability and death worldwide. In 2016, more than 1.9 billion adults were overweight, according to the World Health Organization. According to current projections, by 2030, 60% of the world's population (that is, 3.3 billion people) may be overweight (2.2 billion) or obese (1.1 billion), if trends in obesity continue.

In 2021, the journal Nature Communications published data on the effectiveness of the use of an invasive device that stimulates the efferent fibers of the vagus nerve of the stomach with light fluxes and thereby reduces the severity of hunger. In addition, in small clinical trials in patients with depression and epilepsy treated with transcutaneous vagus nerve stimulation, this procedure has been shown to lead to significant weight loss.

Although the mechanisms are not fully understood, it is believed that a high-calorie diet contributes to the desensitization of the vagus afferent fibers to peripheral signals and leads to a decrease in the constitutive expression of orexigenic receptors and neuropeptides. Violation of signal transmission along the afferent fibers of the vagus nerve may be sufficient for the development of hyperphagia and obesity, and stimulation of the vagus nerve, respectively, can be used in the treatment of these conditions. Recent discoveries revealed a new and important role of the vagus nerve within a physiological mechanism that utilizes afferent and efferent signaling in controlling cytokine levels and inflammation - the inflammatory reflex.

Afferent vagus nerve projections to the GI tract and the hepatic portal system play a major role in communicating alterations in peripheral metabolic homeostasis, including changes in cholecystokinin, lipids, leptin, insulin and glucose levels to the brain. In a reflex manner, efferent vagus nerve innervations of the heart, liver and pancreas provide cardio-metabolic regulatory output. Cholecystokinin- and leptin-induced afferent vagus nerve activity importantly mediates satiety and regulates feeding behavior. Cholecystokinin, released as a result of intestinal lipid accumulation also causes activation of afferent signaling and subsequent efferent vagus nerve output to liver that suppresses hepatic gluconeogenesis.

Transcutaneous vagus nerve stimulation (TENS) involves the stimulation of the left and/or right auricular branch of the vagus nerve in the area of the cymba concha with low-frequency electrical impulses. The auricular branch of the vagus nerve runs superficially, which makes it a favorable target for non-invasive stimulation techniques to modulate vagal activity. It gained popularity due to minimal side effects and low cost.

In recent years, the use of this technology in the treatment of various disorders, including headache, tinnitus, prosocial behavior, atrial fibrillation, associative memory, schizophrenia, traumatic pain, and Crohn's disease, has been explored - chronic conditions characterized by immune and metabolic dysregulation. For this reason, there have been many early-stage clinical trials on a diverse range of conditions. These trials often report conflicting results for the same indication.

In this study, the investigators want to explore: will low-frequency transcutaneous electrical stimulation of the auricular branch of the vagus nerve contribute to weight loss in patients and improve their quality of life?

ELIGIBILITY:
Inclusion Criteria:

Adult patients with grade 1-2 nutritional obesity who are willing and able to give informed written consent to participate in the study, are on sinus rhythm and are not taking any antiarrhythmic drugs, including beta-blockers.

Exclusion Criteria:

* Cardiac arrhythmias: bradyarrhythmias, Atrioventricular blockades of any degree;
* Taking beta blockers;
* The endocrine nature of obesity;
* Expected technical difficulties when using the device on the part of the patient;
* Pregnant or plan on becoming pregnant or breastfeeding during the study period;
* Presence of an electrically, magnetically or mechanically activated implant, an intracerebral vascular clip, or any other electrically sensitive support system.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 131 (Actual)
Dates: Start 2022-04-04 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of body fat | 6-month follow-up
  It is calculated using the body composition analyzer "In Body 910" in dynamics (at the start and at the end of the trial).
Body Mass Index | 6-month follow-up
  BMI will be determined by the equation (kg/m2) in dynamics (at the start and at the end of the trial).
Waist circumference | 6-month follow-up
  Waist circumference will be measured on bare skin midway between the lowest rib and the superior border of the iliac crest using an inelastic measuring tape to the nearest 0.1 cm following the World Health Organization guideline. Measurement will be performed at the start and at the end of the trial.

SECONDARY OUTCOMES:
Total Weight Loss | 6-month follow-up
  The difference in weight in kilograms compared to the baseline value after 6 months observation within the trial.
Percentage of Total Weight Loss | 6-month follow-up
  The ratio of the difference between the weight at the start of the trial and at the end of the trial in relation to the total body weight.
Eating behavior questionnaire | 6-month follow-up
  The investigators will analyse changes in eating behavior using the Food Frequency Questionnaire (FFQ) and the 24-hour replay method.
Hip circumference | 6-month follow-up
  Hip circumference will be taken on bare skin around the widest portion of the buttocks using an inelastic measuring tape to the nearest 0.1 cm and the tape should be placed parallel to the floor.
Waist circumference/Hip circumference | 6-month follow-up
  The ratio of the two values (Waist Circumference/Hip circumference) will be performed at the start and at the end of the trial.
Lean Mass | 6-month follow-up
  Lean mass will be simultaneously determined during the bioimpedance "In Body 910" scan for total body fat mass. Measurement will be performed at the start and at the end of the trial.
Health-related Quality of Life | 6-month follow-up
  The validated short form survey measures health-related quality of life covering physical functioning, emotional and mental health, bodily pain, general health, vitality, and social functioning. A higher overall score indicates better quality of life.
Adherence | 6-month follow-up
  Adherence will be verified by evaluating the completeness of the patient's diary.
Adverse Events | 6-month follow-up
  Adverse events will be closely monitored regularly by research personnel, and by subjects' voluntary reports.

CONTACTS AND LOCATIONS:
Overall Officials: Oxana Drapkina, Principal Investigator — National Medical Research Center for Therapy and Preventive Medicine
Locations (1):
- National Medical Research Center for Therapy and Preventive Medicine, Moscow, Russia

REFERENCES:
- [Background] Kim WS, Hong S, Gamero M, Jeevakumar V, Smithhart CM, Price TJ, Palmiter RD, Campos C, Park SI. Organ-specific, multimodal, wireless optoelectronics for high-throughput phenotyping of peripheral neural pathways. Nat Commun. 2021 Jan 8;12(1):157. doi: 10.1038/s41467-020-20421-8. PMID 33420038
- [Background] Verma N, Mudge JD, Kasole M, Chen RC, Blanz SL, Trevathan JK, Lovett EG, Williams JC, Ludwig KA. Auricular Vagus Neuromodulation-A Systematic Review on Quality of Evidence and Clinical Effects. Front Neurosci. 2021 Apr 30;15:664740. doi: 10.3389/fnins.2021.664740. eCollection 2021. PMID 33994937
- [Background] Stavrakis S, Stoner JA, Humphrey MB, Morris L, Filiberti A, Reynolds JC, Elkholey K, Javed I, Twidale N, Riha P, Varahan S, Scherlag BJ, Jackman WM, Dasari TW, Po SS. TREAT AF (Transcutaneous Electrical Vagus Nerve Stimulation to Suppress Atrial Fibrillation): A Randomized Clinical Trial. JACC Clin Electrophysiol. 2020 Mar;6(3):282-291. doi: 10.1016/j.jacep.2019.11.008. Epub 2020 Jan 29. PMID 32192678
- [Background] Wolf V, Kuhnel A, Teckentrup V, Koenig J, Kroemer NB. Does transcutaneous auricular vagus nerve stimulation affect vagally mediated heart rate variability? A living and interactive Bayesian meta-analysis. Psychophysiology. 2021 Nov;58(11):e13933. doi: 10.1111/psyp.13933. Epub 2021 Sep 2. PMID 34473846
- [Background] Yap JYY, Keatch C, Lambert E, Woods W, Stoddart PR, Kameneva T. Critical Review of Transcutaneous Vagus Nerve Stimulation: Challenges for Translation to Clinical Practice. Front Neurosci. 2020 Apr 28;14:284. doi: 10.3389/fnins.2020.00284. eCollection 2020. PMID 32410932